CLINICAL TRIAL: NCT05536986
Title: Correlation Between Psychological Stress and Progression of Newly Oligodendroglioma Towards Secondary Glioma: A Longitudinal Study Based on Long-term Follow-up
Brief Title: Correlation Between Psychological Stress and Progression of Newly Oligodendroglioma Towards Secondary Glioma
Status: Not yet recruiting | Type: Observational
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HenanPPH-Oligodendroglioma
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Oligodendroglioma, Adult
Keywords: Oligodendroglioma; Psychological stress; progression
MeSH Terms: conditions — Oligodendroglioma; Stress, Psychological; Disease Progression | interventions — Anthropogenic Effects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observation group of newly oligodendroglioma patients with high-level psychological stress: The patients had high threshold levels of perceived psychological stress, fear, anxiety, and depression as assessed by psychologists
  Interventions: Other: Stressors
- Observation group of newly oligodendroglioma patients with low-level psychological stress: The patients had lower than threshold levels of perceived stress, psychological distress, fear, anxiety, and depression as assessed by psychologists

INTERVENTIONS:
Other: Stressors — Patients are exposed to stressful situations related to the diagnosis and treatment of the disease
  Groups: Observation group of newly oligodendroglioma patients with high-level psychological stress

SUMMARY:
It is a single-center, prospective, observational, non-randomized study of newly diagnosed oligodendroglioma patients conducted in a tertiary hospital. The investigators conduct an eight-year follow-up, including patients' psychological stress, immune biomarker changes, quality of life, and disease progression of patients towards secondary glioma after the first definite diagnosis. In the first year after diagnosis, patients are followed up four times at 1 month, 3 months, 6 months, and 12 months. After that, patients are followed up semiannually.

The study had two cohorts, a high-stress cohort and a low-stress cohort, which are grouped after initial recruitment. Both groups undergo total resection of tumors and received 3 months of standardized treatment with radiotherapy and chemotherapy. Neither participants nor doctors but the researcher can choose which group participants are in. No one knows if one study group is better or worse than the other.

DETAILED DESCRIPTION:
Oligodendroglioma belongs to the class of gliomas that represent the most common class of primary malignant human brain tumors in adulthood. After tumor resection, patients still face the possibility of recurrence and even progression to glioblastoma. The immune microenvironment is most likely contributing to their development, but underlying pathomechanisms are only partly understood.

The high-level psychological stress can lead to a change in malignant tumors patients' neuroendocrine pathways and correlates with the prognosis outcome. In addition, psychological stress can lead to changes in the immune microenvironment, but if it leads to disease progression in oligodendroglioma towards secondary glioma has not been adequately demonstrated.

Grouping process: 60 patients are expected to be enrolled. After enrollment, participants will receive regular tumor in situ fluid (fluid within the surgical cavity, TISF) sampling for tumor mutation burden (TMB) analysis and regular MRI. Under the standard of care, participants will receive psychological stress assessment after being diagnosed. according to five psychological scales, and the patients were grouped according to the cut-off value of each scale, the psychological stress of the patients is measured by distress thermometer (DT), perceived stress scale (PSS), anxiety/depression (HADS), and fear of disease progression scale (PoP-Q-SF).

Primary study objectives:

* To evaluate the proportion of patients with tumor recurrence
* To evaluate the changes in immune markers of acute and chronic psychological stress in patients with oligodendroglioma after diagnosis.
* To analyze the classification of recurrent glioma.

Secondary study objectives:

* To evaluate the progression-free survival of patients with different psychological stress levels.
* To evaluate the overall survival of patients with different psychological stress levels.
* To evaluate the quality of life of patients with different psychological stress levels.

Exploratory objectives:

-To evaluate the effect of managing the patient's psychological stress on the patient's immune microenvironment.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* Karnofsky Performance Score ≥ 70 %
* histologically confirmed, previously untreated glioma receiving a standardized chemoradiotherapy regimen
* no previous history of mental illness, drug abuse, or alcohol abuse
* ability to communicate and read and write independently
* willing and able to comply with the protocol as judged by the investigator's signed informed consent.

Exclusion Criteria:

* Patients who have any other disease, either metabolic or psychological, or who have any evidence on clinical examination or special investigations (including laboratory findings) which give reasonable suspicion of a condition that interferes with the adequate measurement of the stress axis (e.g. chronic use of corticosteroids ≥ 3 months before study entry for diseases other than glioblastoma, (dexamethasone use in the context of glioblastoma is allowed) severe, medically treated psychiatric disorder prior to the diagnosis of glioblastoma Participation in a study with investigational drugs.
* pregnancy or breast-feeding
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, neurologic deficits that interfere with the planned walking tests, dementia, or confusional state.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with oligodendroglioma
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-12-20 (Estimated); Primary Completion 2028-12-20 (Estimated); Study Completion 2030-12-20 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with tumor recurrence | From the time of diagnosis to 8 years
  The proportion of patients with oligodendroglioma who had recurrence after tumor resection.
The proportion of patients with high-level psychological stress | From the time of diagnosis to 8 years
  The self-report questionnaire of Perceived Stress Scale (PSS) is used to measure the psychological stress level of patients, with 43 as the critical value, more than or equal to 43 as the high level of psychological stress, less than 43 as the low level of psychological stress.
Tumor mutation burden (TMB) | From the time of diagnosis to 8 years
  The proportion of tumor mutational burden ≥10 Mut/MB in the population who remain progression-free after diagnosis.

SECONDARY OUTCOMES:
The Short Form-36 (SF-36) | From the time of diagnosis to 8 years
  The questionnaire of Short Form-36 (SF-36) is used health-related quality- of-life measure in participants outcomes. The scale contains 9 dimensions with a total score of 100 points.
Progression-free survival at 5 years | From the time of diagnosis to 8 years
  The proportion of participants in the analysis population who remain progression-free for at least 5 years after diagnosis.
Overall survival rate at 8 years | From the time of diagnosis to 8 years
  OS-36 is the proportion of participants in the analysis population who remain alive for at least 8 years after diagnosis.
Progression-free survival at 8 years | From the time of diagnosis to 8 years
  The proportion of participants in the analysis population who remain progression-free for at least 8 years after diagnosis.

OTHER OUTCOMES:
Classification proportion of glioma recurrence | From the time of diagnosis to 8 years
  Patients with recurrent gliomas undergo secondary surgery/needle biopsy to determine the type of recurrent glioma.

CONTACTS AND LOCATIONS:
Overall Officials: Xingyao Bu, Study Director — Henan Provincial People's Hospital

IPD SHARING:
Plan to Share IPD: No